CLINICAL TRIAL: NCT03535532
Title: Effectiveness Comparison of Medical Treatment and Unilateral Laparoscopic Adrenalectomy for Resistant Hypertension in Patients Concomitant With Adrenal Diseases: A Prospective, Multi-Center, Open-Labeled, Randomized Clinical Trial.
Brief Title: Unilateral Laparoscopic Adrenalectomy for Resistant Hypertension in Patients With Adrenal Diseases
Acronym: ULARH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Cai, Director, Hypertension Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULARH2017
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Resistant Hypertension; Adrenal Disease
Keywords: resistant hypertension; Adrenal Disease; medical treatment; laparoscopic adrenalectomy
MeSH Terms: conditions — Adrenal Gland Diseases

STUDY DESIGN:
Intervention Model Description: resistant hypertensive patients diagnosed with adrenal diseases based on imaging tools will be randomly allocated into unilateral laparoscopic adrenalectomy group and standard medical treatment group.
Masking Description: Since one of the intervention is invasive surgical operation, the other is conservative medical treatment, the difference between these two intervention is too obvious to mask, no masking are designed in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unilateral laparoscopic adrenalectomy (Experimental): subjects allocated in this group will be given unilateral laparoscopic adrenalectomy as treatment.
  Interventions: Procedure: unilateral laparoscopic adrenalectomy
- standard medical treatment (Active Comparator): subjects allocated in standard medical treatment group will be given conservative medicine treatment.
  Interventions: Drug: standard medical treatment

INTERVENTIONS:
Procedure: unilateral laparoscopic adrenalectomy — unilateral laparoscopic adrenalectomy is a kind of minimally invasive surgery commonly operated in patients diagnosed with adrenal diseases with a high likelihood of malignance or surplus hormone secretion.
  Other Names: standard medical treatment
  Arms: unilateral laparoscopic adrenalectomy
Drug: standard medical treatment — standard medical treatment: detailed medicine strategy chosen for each patient will be associated with their own conditions based on current guidance recommendations.
  Other Names: unilateral laparoscopic adrenalectomy
  Arms: standard medical treatment

SUMMARY:
ULARH is a 2-arm, prospective, open-labeled, multi-center randomized clinical trial.The purpose of this study is to compare the effectiveness of medical treatment and unilateral laparoscopic adrenalectomy for resistant hypertension in patients diagnosed with adrenal disease based on imaging tools.Relative ratio of end-point events occurence in three years is considered as primary outcome. Furthermore, we will exploit clinical factors which could indicate a favorable outcome in participants who accepted surgical treatment in this study.

DETAILED DESCRIPTION:
Resistant hypertension is a clinical condition characterized by the presence of BP values above the recommended limits of the reference values(BP>140/90 mmHg in hypertensive patients), despite the adherence to appropriate life style changes and to a drug therapy of at least three classes of drugs, one of which is represented by a diuretic, in adequate doses. Several small-sample studies suggest the prevalence of resistant hypertension is about 5-30% in Chinese population. Uncontrolled blood pressure elevation attributes to a higher incidence of stroke, heart failure, chronic renal disease, dementia and cardiovascular deaths. Improving the management of resistant hypertension is a constantly tricky problem in hypertension clinical practice.

Compared with patients whose blood pressure level are more easily to get controlled, patients diagnosed with resistant hypertension presented a higher risk of adrenal anomaly when screened by imaging tools. Current clinical practice guidance recommend unilateral laparoscopic adrenalectomy as a preferable treatment merely for adrenal incidentalomas with over hormone secreting like cortisol or aldosterone, or a high likelihood of malignance. Among patients who meet above surgery indication, the ratio of cure for hypertension varies from approximately 30 to 80%. However, in recent years, there are growing evidence showed that hypertensive patients diagnosed with adrenal disease based on imaging tools also gain much benefit from adrenalectomy even if there is no evidently abnormal hormone secretion. Last year, a prospective cohort study published on <Ann Intern Med> suggested that "nonfunctional" adrenal tumors associate with increased diabetes risk. These studies prompt a re-assessment of the classification of benign adrenal tumors as "non-functional"and their potential damage.

In a retrospective study conducted by our group in early period to evaluate the effect of surgery treatment in resistant hypertensive patients, we found one third of resistant hypertensive patients were cured as well as another one third get improved after unilateral laparoscopic adrenalectomy. Thus, we designed this study, expecting a further and more detailed perception of the relationship between resistant hypertension and adrenal anomaly.

ELIGIBILITY:
Inclusion Criteria:

1. Resistant hypertensive patients diagnosed with adrenal disease based on imaging tools (resistant hypertension defined as the presence of BP values above the recommended limits of the reference values(BP>140/90 mmHg),despite the adherence to appropriate life style changes and to a drug therapy of at least three classes of drugs for at least one month, one of which is represented by a diuretic, in adequate doses)
2. Signed the written informed consent.

Exclusion Criteria:

1. Patients with surgical contraindication;(Performed coronary revascularization (PCI or CABG) within the previous 6 months; Cerebral hemorrhagic stroke within the previous 3 months, or new onset cerebral infarction within the latest 2 weeks;Severe heart failure or kidney disfunction within the previous 6 months)
2. Patients who has proceeded unilateral laparoscopic adrenalectomy once;
3. Severe somatic disease such as cancer;
4. Severe cognitive impairment or mental disorder;
5. Participating in other clinical trials.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-20 (Estimated); Primary Completion 2020-10-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
A composite of end-point events | 3 year
  A composite end-point comprised of myocardial infarction(MI), congestive heart failure, cerebrovascular event, end stage renal disease, death.

SECONDARY OUTCOMES:
Major coronary events | 3 years
  Major coronary events comprised of myocardial infarction (MI), hospitalization for unstable angina or acute decompensated heart failure, coronary revascularization (percutaneous coronary intervention [PCI], coronary artery bypass grafting [CABG]), and death from cardiovascular causes.
First occurrence of symptomatic stroke (ischemic or hemorrhagic, fatal or nonfatal) | 3 years
  First occurrence of symptomatic stroke (ischemic or hemorrhagic, fatal or nonfatal)
All-cause death | 3 years
  All-cause death
Cardiovascular death | 3 years
  Cardiovascular death
myocardial infarction | 3 years
  myocardial infarction
Hospitalization for unstable angina | 3 years
  Hospitalization for unstable angina
Hospitalization for acute decompensated heart failure | 3 years
  Hospitalization for acute decompensated heart failure
coronary revascularization (percutaneous coronary intervention [PCI], coronary bypass grafting [CABG]) | 3 years
  coronary revascularization (percutaneous coronary intervention [PCI], coronary bypass grafting [CABG])
First occurence of diabetes mellitus | 3 years
  First occurence of diabetes mellitus
Decline in cognitive function | 3 years
  Decline in cognitive function includes sensory disturbance, memory disorders and thinking disorders, which is assessed by mini-mental state examination (MMSE)
Decline in renal functio or development of end stage renal disease (ESRD) | 3 years
  Decline in renal function is assessed by any of the following: (1) For patients with chronic kidney disease (eGFR<60 ml per minute per 1.73 m2) at baseline, the renal outcome was a composite of a decrease in the eGFR of 50% or more (confirmed by a subsequent laboratory test) or the development of EDRD requiring long-term dialysis or kidney transplantation; or (2) For participants without chronic kidney disease at baseline, the renal outcome was defined by a decreased in the eGFR of 30% or more to a value of less than 60 ml per minute per 1.73 m2.
Major artery function changes | 3 years
  Major artery function changes are assessed by a composite of decrease in the ankle branchial index [ABI], brachial-ankle pulse wave velocity(baPWV),or brachial artery flow-mediated dilation [FMD].
  ABI and baPWV, well-established non-invasive techniques fr evaluating obstruction and stiffness of peripheral artery respectively, are considered for the purposes of cardiovascular risk assessment. ABI is the ratio of average systolic blood pressure measured in brachial/ankle, and an ABI between and including 0.9 and 1.2 is considered normal, while a lesser than 0.9 indicates arterial disease. The unit measure of baPWV value is cm per second.
  FMD serves as an index of nitric oxide (NO)-mediated endothelium-dependent vasodialator function in humans and is regarded as a surrogate marker of cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, MD, Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (3):
- China (3):
  - Chinese Academy of Medical Sciences, FuWai Hospital, Beijing, Beijing Municipality
  - Shandong Provincial Hospital, Ji'nan, Shandong
  - Yunzhou Municiple Hospital, Ji'ning, Shandong

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet

REFERENCES:
- [Background] Sim JJ, Bhandari SK, Shi J, Reynolds K, Calhoun DA, Kalantar-Zadeh K, Jacobsen SJ. Comparative risk of renal, cardiovascular, and mortality outcomes in controlled, uncontrolled resistant, and nonresistant hypertension. Kidney Int. 2015 Sep;88(3):622-32. doi: 10.1038/ki.2015.142. Epub 2015 May 6. PMID 25945406
- [Background] Lopez D, Luque-Fernandez MA, Steele A, Adler GK, Turchin A, Vaidya A. "Nonfunctional" Adrenal Tumors and the Risk for Incident Diabetes and Cardiovascular Outcomes: A Cohort Study. Ann Intern Med. 2016 Oct 18;165(8):533-542. doi: 10.7326/M16-0547. Epub 2016 Aug 2. PMID 27479926
- [Background] Xu T, Xia L, Wang X, Zhang X, Zhong S, Qin L, Zhang X, Zhu Y, Shen Z. Effectiveness of partial adrenalectomy for concomitant hypertension in patients with nonfunctional adrenal adenoma. Int Urol Nephrol. 2015 Jan;47(1):59-67. doi: 10.1007/s11255-014-0841-8. Epub 2014 Oct 11. PMID 25305227
- [Background] Fassnacht M, Arlt W, Bancos I, Dralle H, Newell-Price J, Sahdev A, Tabarin A, Terzolo M, Tsagarakis S, Dekkers OM. Management of adrenal incidentalomas: European Society of Endocrinology Clinical Practice Guideline in collaboration with the European Network for the Study of Adrenal Tumors. Eur J Endocrinol. 2016 Aug;175(2):G1-G34. doi: 10.1530/EJE-16-0467. PMID 27390021
- [Background] Denolle T, Chamontin B, Doll G, Fauvel JP, Girerd X, Herpin D, Vaisse B, Villeneuve F, Halimi JM. [Management of resistant hypertension. Expert consensus statement from the French Society of Hypertension, an affiliate of the French Society of Cardiology]. Presse Med. 2014 Dec;43(12 Pt 1):1325-31. doi: 10.1016/j.lpm.2014.07.016. Epub 2014 Nov 20. French. PMID 25459067